CLINICAL TRIAL: NCT04903639
Title: Obstructive Sleep Apnea Prevalence in Patients With Chronic Obstructive Pulmonary Diseases
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Marwa Elsayed Elnaggar, Assistant professor of chest diseases, chest department, Faculty of Medicine, Benha University, Benha University
Other Study IDs: BenhaU123
Record Dates: First submitted 2021-05-22; First posted 2021-05-26 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: OSA
Keywords: COPD; OSA; OS; AHI
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obese COPD: COPD patient with BMI more than 30
  Interventions: Diagnostic Test: sleep study
- non obese COPD: COPD patient with BMI less than 30
  Interventions: Diagnostic Test: sleep study

INTERVENTIONS:
Diagnostic Test: sleep study — The polysomnography consists of electroencephalogram (EEG), electrooculogram (EOG), electrocardiogram (ECG), electromyogram (EMG), pulse oximetry, thoracic and abdominal straps, body posture sensor, nasal thermistor and nasal cannula to assess respiratory flow and pressure and bipolar channel limb movements (tibialis anterior). Electrodes and sensors were attached to patients by sleep physiologist. Data collection was obtained following signal perception by preprocessed computer (DOMINO Software, ver. 2.6.0; SOMNO Medics GmbH).

SUMMARY:
The conjunction of chronic obstructive pulmonary disease (COPD) and obstructive sleep apnea (OSA) is known as Overlap Syndrome (OS). The coexistence of these diseases have cardiovascular morbidity and mortality. The aim of this study is to assess the prevalence of OSA in COPD patients. 100 COPD patients (obese and non-obese) performed sleep questionnaires and polysomnogram.

DETAILED DESCRIPTION:
300 patients were enrolled in this prospective observational study who were attended at chest department, outpatient clinic Benha university hospitals for follow up between August 2018 and October 2020. According to medical history, clinical examination and pulmonary function tests, only stable COPD patients (100 patients) were included. The research ethics committee at the faculty of medicine has approved the study and all patients provided informed consent before participation.

COPD patients were divided according to their body mass index (BMI) into two groups ; group A: 50 obese COPD patients (BMI ≥30 kg/m2) and group B: 50 non obese COPD patients (BMI ≤ 29.9 kg/m2).

Inclusion criteria: COPD patients were diagnosed according to the Global initiative for chronic obstructive pulmonary disease on the basis of (GOLD, 2017). Included patients who had chronic cough, sputum production, dyspnea and /or a history of exposure to risk factors for the disease and confirmed by the presence of a post bronchodilator forced expiratory volume in the 1st second/forced vital capacity (FEV1/FVC) < 70% .

Exclusion criteria included patients with COPD exacerbation, patients with decompensated heart failure, thyroid dysfunction, ears, nose and throat (ENT) causes of OSA or patients with impaired hepatic and renal function.

COPD patients were characterized by their postbronchodilator FEV1 into mild (FEV1 ≥ 80% anticipated), moderate (50%≤FEV1 < 80% anticipated) and severe (30%≤FEV1 < 50% anticipated).

All patients included in this study were subjected to full history taking, physical examination (general including BMI and neck circumference (NC), local chest examination, oral and ENT), questionnaires [The Epworth Sleepiness Scale (ESS) which translated to Arabic, STOP-Bang Questionnair (SBQ), modified medical research council (mMRC) breathlessness scale which was translated ta Arabic, spirometry which was done using JAEGER carefusion Germany 234 GmbH Lelbnizstr .7, 97204 Hoechberg, Germany. Spirometry was done during stability of the disease. Echocardiography, liver, kidney and thyroid function tests were done .Overnight Polysomnography (PSG) (SOMNO Screen Plus; SOMNO Medics GmbH, Randersacker, Germany). The polysomnography consists of electroencephalogram (EEG), electrooculogram (EOG), electrocardiogram (ECG), electromyogram (EMG), pulse oximetry, thoracic and abdominal straps, body posture sensor, nasal thermistor and nasal cannula to assess respiratory flow and pressure and bipolar channel limb movements (tibialis anterior). Electrodes and sensors were attached to patients by sleep physiologist. Data collection was obtained following signal perception by preprocessed computer (DOMINO Software, ver. 2.6.0; SOMNO Medics GmbH).

Patients considered having OSA if they had apneic episodes occurred in the existence of respiratory muscle effort and lasted 10 seconds or more, or have a combination of apneas and hypopneas. The apnea-hypopnea index (AHI) is gotten from the absolute number of apneas and hypopneas separated by the total sleep time. Cutoff levels on AHI incorporate 5-15 episodes per hour for mild, 15-30 episodes per hour for moderate and more than 30 episodes per hour for severe OSA

ELIGIBILITY:
Inclusion Criteria:

• stable COPD patients

Exclusion Criteria:

* patients with COPD exacerbation
* patients with decompensated heart failure
* patients with thyroid dysfunction
* ears, nose and throat (ENT) causes of OSA
* patients with impaired hepatic and renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who had chronic cough, sputum production, dyspnea and /or a history of exposure to risk factors for the disease and confirmed by the presence of a post bronchodilator forced expiratory volume in the 1st second/forced vital capacity (FEV1/FVC) < 70%. COPD patients were characterized by their postbronchodilator FEV1 into mild (FEV1 ≥ 80% anticipated), moderate (50%≤FEV1 < 80% anticipated) and severe (30%≤FEV1 < 50% anticipated).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
prevalence of OSA in COPD patients | through study completion, an average of 1 year
  number of AHI found during sleep study of COPD patients
prevalence of OSA in COPD patients | through study completion
  number of AHI found during sleep study of COPD patients

CONTACTS AND LOCATIONS:
Overall Officials: M E Elnaggar, MD, Principal Investigator — Assistant professor of chest diseases, Faculty of Medicine, Benha University
Locations (1):
- Faculty of medicine, Benha University, Banhā, Alqalubia, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD could be shared depending on personal request